CLINICAL TRIAL: NCT01479738
Title: The Second Hospital of Qinhuangdao, Qinhuangdao, Hebei, 066600, China
Brief Title: Proximal Interphalangeal Joint Arthroplasty Using a Graft From the Capitate
Acronym: PIPPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Qinhuangdao (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: SHQ002
Record Dates: First submitted 2011-11-19; First posted 2011-11-24 (Estimated); Last update posted 2011-11-28 (Estimated); Status verified 2011-11

CONDITIONS: Recurrent Dislocation of Hand
Keywords: arthroplasty; graft; capitate; artery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Capitate bone grafting (Experimental): 18 patients with PIP joint defects were included in the study. There were 13 male and 5 female patients with a mean age of 31 years (range, 18-47 years). The injury occurred in the right hand in 11 patients and on the left hand in 7. The injured PIP joints were in the index finger (n=7), long finger (n=9), and ring finger (n=2).
  Interventions: Procedure: Capitate bone grafting

INTERVENTIONS:
Procedure: Capitate bone grafting — Capitate bone graft transfer for PIP joint reconstruction

SUMMARY:
The capitate had a widened distal base. The distal articulation can be used for proximal interphalangeal (PIP) articula reconstruction.

DETAILED DESCRIPTION:
Previous anatomical studies have shown that the capitate had a widened distal base. The distal articulation was mainly with the base of the third metacarpal and partially with the base of the second metacarpal. The articulation was slightly flattened with a convex and concave dorsal articular surface. The contour stimulates our imagination and creativity to use a portion of the articular surface for PIP arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

1. an articular defect at the proximal aspect of the PIP joint;
2. the defect larger than 5 mm × 5 mm in size based on intraoperative findings.

Exclusion Criteria:

1. large defects involved double joint surfaces;
2. the size of the defect less than 5 mm × 5 mm;
3. mult-digital articular defects that all required osteoarticular grafting;
4. associate with infection or other diseases that restrict to use the technique.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2005-01; Primary Completion 2011-08 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
range of motion | 37 to 46 months postoperatively
  Active range of motion of the hand were measured by a goniometer.

SECONDARY OUTCOMES:
grip strength | 37 to 46 months postoperatively
  The grip strength of the thumb to the injured finger was measured using dynamometers
pinch strength | 37 to 46 months postoperatively
  The pinch strength of the thumb to the injured finger was measured using dynamometers

CONTACTS AND LOCATIONS:
Overall Officials: Xu Zhang, M.D., Study Chair — The Second Hospital of Qinhuangdao
Locations (1):
- The second hospital of Qinhuangdao, Qinhuangdao, Hebei, China

REFERENCES:
- [Background] Freiberg A. Management of proximal interphalangeal joint injuries. Can J Plast Surg. 2007 Winter;15(4):199-203. doi: 10.1177/229255030701500407. PMID 19554177
- See also: Management of proximal interphalangeal joint injuries — http://www.ncbi.nlm.nih.gov/pubmed/19554177